CLINICAL TRIAL: NCT07369687
Title: Parent-administered Pediatric Tuina With Routine Care Versus Routine Care Alone for Pediatric Functional Dyspepsia: a Pilot Randomized Controlled Trial
Brief Title: Parent-administered Pediatric Tuina Versus Routine Care for Pediatric Functional Dyspepsia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT_PFD_AS
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Functional Dyspepsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: parent-administered pediatric tuina (n=25) (Experimental)
  Interventions: Other: parent-administered pediatric tuina
- Control group: routine care (n=25) (No Intervention)

INTERVENTIONS:
Other: parent-administered pediatric tuina — Parents in parent-administered pediatric tuina group will attend an online training session (within 2 hours) on pediatric tuina for PFD by Hong Kong registered Chinese medicine practitioners and their children will receive 1st TCM pattern identification with 1st individualized pediatric tuina prescription at Baseline. In Week 4, the participant's children will receive the 2nd TCM pattern identification (the 2nd individualized pediatric tuina prescription and the according manipulation trainings will be provided). Parents are also required to deliver 30-minutes pediatric tuina on their child every other days during the 8 week-study period.
  Arms: Intervention group: parent-administered pediatric tuina (n=25)

SUMMARY:
Title: Parent-administered pediatric tuina with routine care versus routine care alone for pediatric functional dyspepsia: a pilot randomized controlled trial Background: Pediatric functional dyspepsia (PFD) is a common gastrointestinal disorder in children, characterized by chronic or recurrent upper abdominal discomfort without identifiable organic causes. Despite education, dietary, and pharmacological interventions, treatment outcomes remain suboptimal. Traditional Chinese Medicine (TCM) pediatric tuina, a specialized massage therapy specifically for children, has shown promise as a complementary approach, including when administered by parents at home; however, evidence regarding its feasibility and effectiveness is still limited.

Objectives: This study aims to evaluate the feasibility, acceptability, and preliminary effects of parent-administered pediatric tuina (PPT) for children with PFD.

Hypothesis: Children receiving PPT will experience greater improvements in PFD symptoms, eating behavior, sleep quality, and quality of life compared to those receiving routine care (RC) over an 8-week period.

Design and subjects: This is a pilot randomized controlled trial involving 50 parent-child dyads (children aged 3-7 years with PFD) recruited from the community. Participants will be randomized into a PPT group or an RC group at 1:1 ratio.

Interventions: Parents in the PPT group will attend two 2-hour training sessions delivered by a registered TCM practitioner to learn the principles and techniques of pediatric tuina. They will administer pediatric tuina sessions (30 minutes every two days) at home for 8 weeks, tailored to their child's specific TCM diagnosis. The RC group will continue their usual care without additional interventions during the study period.

Main outcome measures: The primary outcome measure is the Questionnaire on Pediatric Gastrointestinal Symptoms-Rome IV (QPGS-RIV) to assess PFD symptoms. Secondary measures include eating behavior (Children's Eating Behavior Questionnaire), sleep quality (Sleep Disturbance Scale for Children), quality of life (Pediatric Quality of Life Inventory), and parental stress (Parenting Stress Index-Short Form). Outcome assessment will be conducted at baseline, week 4, and week 8. Acceptability, feasibility, satisfaction, adherence, and safety of the intervention will also be assessed.

Data analysis: A linear mixed-effects model will be employed to analyze group-by-time interactions for all outcomes. Adherence and acceptability will be described qualitatively and quantitatively. Statistical significance is set at p < .05. Thematic analysis will be conducted for qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for the children are the following:

  1. age 3-7 years, which represents the optimal period for both pediatric tuina effectiveness and TCM syndrome differentiation for PFD intervention.
  2. documented PFD diagnosis based on ROME IV criteria.
* Inclusion criteria for the parents are the following:

  1. ability to communicate in Cantonese or Mandarin.
  2. willingness to learn and practice intervention techniques
  3. availability to attend training sessions at The Hong Kong Polytechnic University.
  4. signed informed consent.

Exclusion Criteria:

* Exclusion criteria for the children are the following:

  1. current receipt of tuina or massage treatments.
  2. concurrent acute infectious diseases (scarlet fever, chickenpox), hemorrhagic diseases, skin conditions (burns, severe skin lesions, infections), or severe conditions contraindicated for pediatric tuina (fractures, paraplegia).
* Exclusion criteria for the parents are the following:

  1. severe psychiatric disorders (e.g., major depression) or physical conditions hindering intervention delivery.
  2. Montreal Cognitive Assessment (MoCA) score <22 points.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-04-26 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
The Questionnaire on Pediatric Gastrointestinal Symptoms-Rome IV (QPGS-RIV) Chinese version | Baseline, week 4, and week 8
  The Questionnaire on Pediatric Gastrointestinal Symptoms-Rome IV (QPGS-RIV) is a standardized parent-report measure designed to assess gastrointestinal symptoms in children according to Rome diagnostic criteria. The parent-reported questionnaire evaluates multiple domains including abdominal pain/discomfort, bowel habits, eating patterns, and associated symptoms.

SECONDARY OUTCOMES:
Daily defecation diary Chinese version | Baseline, week 4, and week 8
  Daily defecation diary will document stool frequency, consistency (Bristol stool form scale), straining, toileting time, and soiling episodes throughout the intervention and follow-up periods.
The Children's Eating Behavior Questionnaire (CEBQ) Chinese version | Baseline, week 4, and week 8
  The Children's Eating Behavior Questionnaire (CEBQ) is a 35-item parent-report measure questionnaire assessing eating style in children. Eating style is assessed on eight scales: food responsiveness (4 items), enjoyment of food (4 items), emotional overeating (4 items), desire to drink (3 items), satiety responsiveness (5 items), slowness in eating (4 items), and emotional undereating (4 items), and fussiness (7 items). Informants rate the frequency of their child's behaviors and experiences on a 5-point scale: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always.
The Sleep Disturbance Scale for Children (SDSC) Chinese version | Baseline, week 4, and week 8
  The Sleep Disturbance Scale for Children (SDSC) is a 26-item parent-report questionnaire that evaluates children's sleep problems, assessing children's sleep problems across 6 domains: disorders of initiating and maintaining sleep, sleep breathing disorders, disorders of arousal, sleep-wake transition disorders, disorders of excessive somnolence, and sleep hyperhidrosis. Each item is scored on a 5-point Likert scale from 1-5. The higher the total score, the more serious the sleep disturbance is, and a total score of more than 39 is considered to be a sleep disturbance.
The Pediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL) Chinese version | Baseline, week 4, and week 8
  The Pediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL) is a 23-item parent-report measure of children's health-related quality of life across 4 domains: physical, emotional, social, and school functioning. Parents rate each item on a 5-point scale from 0 (never a problem) to 4 (almost always a problem). Domain scores are computed by transforming items to a 0-100 scale with higher scores indicating better quality of life.
The Parenting Stress Index-Short Form (PSI-SF) Chinese version | Baseline, week 4, and week 8
  The Parenting Stress Index-Short Form (PSI-SF) is a 36-item self-report measure assessing parental stress levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No